CLINICAL TRIAL: NCT06523218
Title: A Clinical Trial to Investigate the Efficacy of a Supplement to Improve and Maintain Cognitive Function and Memory
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scale Media Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20429
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Decline; Cognitive Function
Keywords: Cognitive Health; Healthy Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MindMD Supplement (Experimental): Participants in the experimental group will receive the MindMD supplement, which contains the following ingredients: 600 mg Bacopa monnieri (Bacognize®), 250 mg Cognigrape® Grape Extract, 100 mg Phosphatidylserine, 50 mg Green Tea Leaf Extract, 1.7 mg Vitamin B6, and 200 mcg Folate (120 mcg folic acid).
  Interventions: Dietary Supplement: MindMD Supplement
- Placebo (Placebo Comparator): Participants in the placebo group will receive a placebo, which contains rice flour encapsulated in a vegetable cellulose capsule.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MindMD Supplement — Participants will take two capsules of the MindMD supplement once daily with their morning meal for a duration of 3 months. The supplement is designed to improve and maintain cognitive function and memory.
  Arms: MindMD Supplement
Other: Placebo — Participants will take two capsules of the placebo once daily with their morning meal for a duration of 3 months. The placebo is designed to be indistinguishable in appearance and administration from the MindMD supplement to ensure blinding.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of 1MD Nutrition's MindMD supplement in improving and maintaining cognitive function and memory. The randomized controlled trial will include 50 healthy participants aged 50-75 years, lasting for 3 months. Participants will be randomized to receive either the test product or a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years
* Regular experience of symptoms related to cognitive decline (e.g., forgetfulness, lack of focus, brain fog)
* Generally healthy without uncontrolled chronic diseases
* Willingness to avoid certain medications and supplements during the study

Exclusion Criteria:

* Any medical condition or treatment impacting cognitive ability Mental health or neurological disorders
* Severe allergies, particularly to soy or other product ingredients
* Taking blood thinning medication
* Recent or planned surgeries
* Major illness in the past three months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-08-17 (Estimated); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function and Memory Improvement | Baseline, Month 2, and Month 3
  Measurement of cognitive function and memory through Cognitive Battery Testing. The Cognitive Battery Testing includes assessments such as Polygons, Double Trouble, Feature Match, Paired Associates, Digit Span, and Spatial Planning. These assessments provide objective measurements of various cognitive functions, including processing speed, memory recall, selective attention, and executive function.

SECONDARY OUTCOMES:
Participants' Perceptions of Cognitive Function and Memory using the Cognitive Function Questionnaire | Baseline, Month 1, Month 2, and Month 3
  Evaluation of participants' self-reported perceptions of the effect of the MindMD supplement on cognitive function and memory. This includes aspects such as focus and attentiveness, comprehension and mental clarity, learning acuity, absentmindedness, and overall quality of life. These perceptions will be measured through the Cognitive Function Questionnaire (CFQ) at specified time points: Baseline (Day 0), Month 1, Month 2, and Month 3.
Participants' Quality of Life | Baseline, Month 1, Month 2, and Month 3
  Assessment of participants' quality of life using the WHO-5 Well-Being Index. These assessments will be conducted at Baseline (Day 0), Month 1, Month 2, and Month 3.
Participants' Focus and Attentiveness | Baseline, Month 1, Month 2, and Month 3
  Evaluation of participants' focus and attentiveness using the Visual Analog Scale (VAS). These assessments will be conducted at Baseline (Day 0), Month 1, Month 2, and Month 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No